CLINICAL TRIAL: NCT02562365
Title: A Phase II,Randomized Study of Adjuvant Chemotherapy of Three-step Regimens (ACTS) in Stage IIIc and Stage IV Epithelial Ovarian, Fallopian Tube, and Primary Peritoneal Cancer (EOC, FTC, PPC)
Brief Title: Adjuvant Chemotherapy of Three-step Regimen in Ovarian Cancer
Acronym: ACTS
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Xiaohua Wu MD (Other)
Responsible Party: Sponsor-Investigator, Xiaohua Wu MD, Fudan University Shanghai cancer center, Fudan University
Organization: Fudan University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: FUSCC-OC1501
Record Dates: First submitted 2015-09-27; First posted 2015-09-29 (Estimated); Last update posted 2022-07-27 (Actual); Status verified 2022-07

CONDITIONS: Ovarian Cancer
Keywords: adjuvent chemotherapy; ovarian cancer
MeSH Terms: conditions — Ovarian Neoplasms | interventions — Etoposide; Cyclophosphamide; Carboplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- A: three steps chemotherapy (Experimental): Cyclophosphamide 400mg（250mg/m2）+Etoposide 100mg (70mg/m2)d1-d3 iv 4w/6cycles , followed by Carboplatin (AUC=5)+Cyclophosphamide 600mg(400mg/m2)d1-d2 iv 8w/6cycles.
  Interventions: Drug: Etoposide, Cyclophosphamide, Carboplatin
- B: Follow-up (No Intervention): No interevention

INTERVENTIONS:
Drug: Etoposide, Cyclophosphamide, Carboplatin — CTX 400mg（250mg/m2）+VP-16 100mg (70mg/m2)d1-d3 iv 4w/6cycles , CBP(AUC=5)+CTX 600mg(400mg/m2)d1-d2 iv 8w/6cycles
  Other Names: VP-16,CTX,CBP
  Arms: A: three steps chemotherapy

SUMMARY:
Ovarian cancer was mostly diagnosed at late stage (III/IV) with high rate of recurrence after first line of therapy by optimal cytoreductive sugery and 6-8cycle of TP chemotherapy. We developed an adjuvant chemotherapy of "three steps" (ACTS). It is adding CTX+VP-16(second step)6cycle and CTX+CBP(third steps) to firstline chemotherapy (first step). The aim of this study is to verify the effectivity and safety of ACTS.

DETAILED DESCRIPTION:
More than 70 percent of ovarian cancer patients were diagnosed in the advanced stage. Currently the 5-year disease free survival (DFS) of stageⅢC-Ⅳovarian cancer patients was about 10 percent after first line chemotherapy. Dr Cai shumo developed adjuvant chemotherapy of "three steps" (ACTS) for advanced ovarian cancer after cytoreductive surgery, based on his 60+ years experience on gynecologic oncology. After the first step 6-8 cycle paclitaxel plus carboplatin chemotherapy, the chemo-sensative cancer cells were killed, but resistant/dormancy cell remained. The second step chemotherapy which is 6 cycle CTX+VP-16 every 4weeks, using different mechanism to kill cancer cells, may decrease the rate of recurrence within 6 month after first step chemotherapy, prolong platinum-free duration and also with acceptable side effects. After second step chemotherapy, in absence of 6 months platinum treatment, the previous G0 dormancy cell may become flexible to platinum treatment. Therefore, in the third step chemotherapy, CTX+CBP is used in every 8 week for 6 cycles. Comparing to using targeted therapy for maintaining therapy, the ACTS cost less.

In the previous observation study(CHINA ONCOLOGY 2013 Vol.23 No.12 p980), In study arm A, the patients received three-step chemotherapy after primary debulking surgery, step one with paclitaxel plus carboplatin (TC regimen), every 3 weeks for 6 to 8 cycles; step two with etoposide plus cyclophosphamide, every 4 weeks for 6 cycles; step three with carboplatin plus cyclophosphamide every eight weeks for six cycles. In control arm B, investigators retrospectively analysed 51 cases withⅢC-Ⅳstage ovarian cancer, who had completely response after standard chemotherapy with six to eight cycles of TC after primary surgery during 2007. Investigators compared the 5-year DFS between the two arms. Results: The 5-year DFS of 15 cases in arm A was 80%(12/15), which was signiifcantly higher than that of arm B (5.9%, 3/51, P<0.01). Therefore we start this randomized open control clinic trial to evaluated the effect of ACTS on overall survival and its safety.

ELIGIBILITY:
Inclusion Criteria:

* Female patients 18-70 years of age.
* ECOG 0-2
* Histologically-confirmed epithelial ovarian or fallopian-tube cancer or primary peritoneal cancer
* FIGO2014 stage IIIC/IV,
* Patients should have received optimal cytoreductive surgery with residual tumor ≤ 1cm and no more than 9 cycle paclitaxel + platinum chemotherapy achieved complete remission (accessed ) and normal CA125.
* No more than 8 months after the last chemotherapy.
* Adequate bone marrow and hepatic function at Screening:

  * Hemoglobin ≥9 g/dL
  * White blood cell count ≥3.0 × 109/L
  * Absolute neutrophil count ≥1.5 × 109/L
  * Platelet count ≥100 × 109/L
  * AST (SGOT)/ALT (SGPT) ≤2.5 ULN
  * Bilirubin <1.5 × ULN
  * Creatinine <1.5 × ULN.
* Ability and willingness to give written informed consent.

Exclusion Criteria:

* Primary or secondary immune deficiency.
* Any uncontrolled medical condition that may put the patient at high risk during treatment .
* Receipt of any other investigational medicinal product within the last 30 days before randomization.
* Patients with second primary cancer, except: adequately treated non-melanoma skin cancer, curatively treated in-situ cancer of the cervix, Ductal Carcinoma in Situ (DCIS), stage 1 grade 1 endometrial carcinoma, or other solid tumors including lymphomas (without bone marrow involvement) curatively treated with no evidence of disease for ≥ 5 years.
* Severe heart/ lung/ liver/ kidney failure.
* uncontroled or active infection disease.
* Legal incompetence, limited legal competence, or detainment in an institution for official or legal reasons.
* Receipt of pelvic or abdominal radiotherapy
* Mucinous adenocarcinoma,clear cell carcinoma, low grade carcinoma

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 130 (Estimated)
Dates: Start 2015-11; Primary Completion 2023-11 (Estimated); Study Completion 2023-11 (Estimated)

PRIMARY OUTCOMES:
overall survival | 5 year

SECONDARY OUTCOMES:
Progression-Free-Survival | 5 year
Health-related quality of life | 5 year
  FACT-O 4.0

CONTACTS AND LOCATIONS:
Overall Officials: Xiaohua WU, PhD & MD, Principal Investigator — Fudan university shanghai cancer center, Deparment of gynecologic oncology
Locations (1):
- Wu Xiaohua, Shanghai, Shanghai Municipality, China

REFERENCES:
- [Derived] Zheng Z, Wang H, Yang H, Tang J, Cheng X, Zhang M, Ren Y, Chen X, Ju X, Xu L, Wu X. Efficacy of Maintenance Therapy With Adjuvant Chemotherapy of Three Steps in Patients Newly Diagnosed With Advanced Ovarian Cancer: A Phase II Randomised Clinical Trial. BJOG. 2025 Jun;132(Suppl 4):52-61. doi: 10.1111/1471-0528.18178. Epub 2025 Apr 28. PMID 40292604